CLINICAL TRIAL: NCT03612102
Title: Evaluating Intensive Group Behavioral Treatment for Children With Selective Mutism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); American Psychological Association (APA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 800008139
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Selective Mutism
Keywords: Selective Mutism; Treatment; Anxiety; Intensive Treatment; CBT; Group Treatment
MeSH Terms: conditions — Mutism; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Families of children with selective mutism will be randomly assigned to receive either immediate intensive group behavioral treatment (IGBT) or to a waitlist with psychoeducational materials, and then IGBT.
Who Masked: Outcomes Assessor
Masking Description: "Independent evaluators" assigned to assess outcomes will be masked to whether or not families participated in IGBT or were at the end of their waitlist period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): The treatment consists of a 5-day intensive group behavioral treatment program (IGBT)
  Interventions: Behavioral: Intensive Group Behavioral Treatment (IGBT)
- Waitlist (No Intervention): The waitlist consists of a 4-week waitlist period where parents will be provided with psychoeducational materials about their child's condition (i.e., selective mutism). After the 4-week waitlist period, families will be provided with the opportunity to participate in IGBT.

INTERVENTIONS:
Behavioral: Intensive Group Behavioral Treatment (IGBT) — IGBT is a 5-day intensive treatment program, where cognitive behavioral therapy is provided to children and their parents delivered over 6-8 hours per day over the course of 5 days.
  Arms: Treatment

SUMMARY:
This goal of this study is to evaluate an intensive group behavioral treatment (IGBT) program for children with selective mutism, a low base-rate childhood anxiety disorder. 29 children between the ages of 5 and 9 will be randomly assigned to participate in a 5-day IGBT over the summer or to a waitlist control condition, with the opportunity to participate in IGBT 4 weeks later. All children that participate in treatment will be followed up 8 weeks into the following school year.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for selective mutism
* Verbal with at least 1 parent or caregiver
* Child fluent in English

Exclusion Criteria:

* Any mental health difficulty significantly more impairing than selective mutism

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions Scales - Improvement (CGI-I) | 5 minutes
  CGI-I is the most widely used clinician-rated measure of treatment-related changes in functioning (Guy & Bonato, 1970) and will be completed by masked independent evaluators in the present study. The CGI-I rates clinical improvement on a 7-point scale, ranging from 1 ("very much improved") to 7 ("very much worse").

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule for Children (ADIS) | 2 hours
  The ADIS is is a semi-structured diagnostic interview that assesses child psychopathology in accordance with DSM criteria. From the ADIS, clinical severity ratings are generated by independent evaluators (IEs) to determine severity of selective mutism and social anxiety disorder. IE's also determine presence of diagnosis, which was also a main outcome.
Selective Mutism Questionnaire (SMQ) | 10 minutes
  The SMQ is a parent-report measure of selective mutism/verbal behaviors in various settings. Two subscales were used for the purpose of this study, the "Social" subscale ("social" scores are a sum of 5 items with scores ranging from 0-15) and the "Home" subscale ("home" scores are a sum of 6 items with scores ranging from 0-18). Lower scores indicate less verbal behavior, and higher scores indicate more verbal behavior.
Children's Global Assessment Scale (CGAS) | 5 minutes
  The Children's Global Assessment Scale (CGAS; Shaffer et al., 1983) is a widely used measure of overall child disturbance, providing a clinician-rated index of functioning. Scores range from 0-100, with lower scores indicating greater functional impairments.
Child Behavior Checklist (CBCL) | 30 minutes
  The CBCL is a parent-report general measure assessing multiple problems of childhood. Subscales are standardized by age and gender. The "Anxiety Problems" Subscale t-score will be used as an outcome measure for the purpose of this study.
School Speech Questionnaire (SSQ) | 5 minutes
  The SSQ is a brief measure given to teachers to assess verbal behavior in the school setting. The SSQ generates a total score, which is a sum of 7 items. Scores range from 0-21, with lower scores indicating less verbal behavior, and higher scores indicating more verbal behavior.
Impairment Rating Scale (IRS) | 8 minutes
  The IRS is a brief teacher-report scale of how much a child's "problems" are interfering with their social and academic functioning in the school setting. The IRS consists of 7 items, with 6 of the items being rated on a scale from 0-6, with higher scores being more indicative of a worst problem. The 6 items are summed to form a total score which ranges from 0 to 36, with higher scores indicating worse problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided